CLINICAL TRIAL: NCT04152785
Title: Measurement of Greenhouse Gas Emissions From Meals of a University Food Operator
Acronym: Cafeteria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Ministère de l'environnement et lutte contre les changements climatiques (Unknown)
Responsible Party: Principal Investigator, Véronique Provencher, Researcher, Laval University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: to be determined
Record Dates: First submitted 2019-10-28; First posted 2019-11-05 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Food Selection
Keywords: environmental concerns; nutrient profiling
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GHG (Experimental): Information given regarding greenhouse gas emissions via a GHG score
  Interventions: Behavioral: Information regarding GHG and/or nutrition
- Nutrition (Experimental): Information given regarding nutrition via a nutrient profiling score
  Interventions: Behavioral: Information regarding GHG and/or nutrition
- GHG+nutrition (Experimental): Information given regarding GHG and nutrition via a combined score
  Interventions: Behavioral: Information regarding GHG and/or nutrition
- No logo (Placebo Comparator): No information given
  Interventions: Behavioral: Information regarding GHG and/or nutrition

INTERVENTIONS:
Behavioral: Information regarding GHG and/or nutrition — Participants will have to select a meal from a menu.

SUMMARY:
Université Laval wishes to raise awareness among students and employees in the university community so that they become aware of the impacts of their consumption choices by equipping them to adopt consumption behaviours that are favourable to the environment and their health. To do this, it is necessary to assess consumers' perception of the information available when choosing a meal to determine, among other things, whether knowledge of greenhouse gas (GHG) emissions influences their selections. In addition to this evaluation criterion, consumer perception of the nutritional quality of food will also be assessed. The nutritional composition of the meals of the characterized week will make it possible to calculate, using a nutritional profiling tool, the nutritional quality score of each meal of the day.

DETAILED DESCRIPTION:
This study consists of an individual meeting with each participant. This meeting will last approximately 1 hour during which each subject will choose a meal and complete various questionnaires. Subjects (male or female) will be randomly assigned to one of the four experimental conditions ("GHG", "nutrition", "GHG+nutrition" and "no logo"). Since subjects could change their eating behaviours if they knew the true purpose of the study, they will be deliberately misled when they enter the study. Participants will be recruited to participate in a market research study in which they will be invited to taste and evaluate a new meal for the cafeteria. At the end of the session, each participant will be informed of the actual objective of the study.

In this context, the general objectives of this second phase of the project are therefore:

1. Evaluate consumer perceptions of the available information on the GHG score (in equivalent C02), the nutritional quality score and the eco-efficiency score (combination of GHG + nutrition), and;
2. Determine if the presence of information (logo on the different scores) influences food choice and consumption among Université Laval students and staff.

ELIGIBILITY:
Inclusion Criteria:

* Study or work at Université Laval

Exclusion Criteria:

* People taking drugs that may affect appetite (e.g., antidepressants, antipsychotics or corticosteroids);
* People with food allergies or intolerances, and pregnant and lactating women;
* People with food aversions to more than 20% of the main meal ingredients from the menu.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — We would like to recuit an equal number of women and men.
Enrollment: 160 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Consumer perceptions of the meal given the information available on the GHG score, the nutritional quality score and the eco-efficiency score (combination of GHG + nutrition) vs no logo. | Within the year after the beginning of the study
  Visual analogue scale (150mm) evaluating the perception of the participants according to the information given. Participants draw a line on the scale (between 0 and 150 mm). The higher the score, the higher the appreciation.

SECONDARY OUTCOMES:
Food choice by the students and staff at Université Laval depending on the presence of information (logo on the different scores). | Within the year after the beginning of the study
  Which meal between the 2 meals presented will be chosen by the participants given the information (logos or no logo) they received.
Amount of the meal consumed by the students and staff at Université Laval depending on the presence of information (logo on the different scores). | Within the year after the beginning of the study
  Measured in grams of food before and after the meal.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Nutraceuticals and Functionnal Foods (INAF), Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No